CLINICAL TRIAL: NCT02134587
Title: Implementation of a Hospital Pharmacovigilance Service and Comparison of Algorithms for Adverse Drug Reaction Causality Assessment
Brief Title: Educational Intervention in Pharmacovigilance for Hospital Health Professionals
Acronym: EIPhv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Fabiana Rossi Varallo, Clinical pharmacist and PhD student, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E015/10
Record Dates: First submitted 2014-05-05; First posted 2014-05-09 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Adverse Drug Reaction
Keywords: Health knowledge, attitudes, practices.; Adverse drug reaction reporting systems.; Pharmacovigilance. Product Surveillance, Postmarketing.; Drug-related side effects and adverse reactions.
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects post educational intervention (Other): Multifaceted educational intervention in pharmacovigilance
  Interventions: Other: Multifaceted educational intervention

INTERVENTIONS:
Other: Multifaceted educational intervention — 1. Application of questionnaire of knowledge, attitudes and skills in pharmacovigilance.
  2. Lecture regarding the theoretical framework and importance of pharmacovigilance, and distribution of educational material
  3. Distribution of educational material
  4. Practical class to explain the correct fill of adverse drug events form
  5. Reapplication of questionnaire of knowledge, attitudes and skills in pharmacovigilance.

SUMMARY:
Spontaneous reports by health professionals generate the signals in pharmacovigilance. However, the passive method has limitations and the most important of them are the underreporting and the poor quality of data, hindering the causality assessment of adverse drug events (ADE). Therefore, the present study aimed to validate an educational intervention (EI) in pharmacovigilance for hospital health professionals, in order to analyze the impact on the knowledge, skill and attitude in ADE reporting.

Investigators proposed a multifaceted EI which will be developed in four meetings with one hour each. The following activities will be carried out: application of a questionnaire to assess the knowledge, skill and attitude before and after EI; lecture; practical class and education material distribution. The answers of questionnaire are going to be analyzed using content analysis technique. The definitions of World Health Organization and the minimum and desired criteria to fill the ADE form, according to the Pan American Health Organization, are going to be considered gold-standard answers. The statistical test of Wilcoxon-Mann Whitney test for paired samples will be applied, in order to assess the impact of educational intervention on behavior of health professionals (ADE reporting).

With the present study, the following hypotheses will be tested:

H0= There is no difference between the numbers of ADE reported (behavior/attitudes) before and after the educational intervention.

H1= The numbers of ADE reported before and after the educational intervention are different.

DETAILED DESCRIPTION:
A quasi-experimental study with health professionals who acted in a general and public hospital of medium complexity with 104 beds will be performed.

Investigators proposed an educational intervention, with the development of lecture and practical class, application of questionnaire before and after EI and the distribution of educational material. Activities will be developed in four meetings of one hour each one.

In the first meeting, questionnaire will be applied, in order to assess knowledge, skills and attitudes in pharmacovigilance prior to EI. The instrument was elaborated based on previous studies. Second meeting will be comprise a lecture regarding the theoretical framework and importance of pharmacovigilance, and distribution of educational material, whose content includes the same issues of presentation. In the third meeting, a practical class will be performed to promote a discussion of a fictitious case of adverse drug reaction (ADR), in order to elucidate the correct fill of ADE form. In the fourth meeting, will be repeated the application of questionnaire, in order to assess the impact of EI. With the aim to verify change behavior of health professionals regarding pharmacovigilance activities, the number of ADE reports made prior and after intervention will be compared.

ELIGIBILITY:
Inclusion Criteria:

All health professionals (physicians, pharmacists, nurses, auxiliaries of nurses and pharmacists, as well as the multidisciplinary team - social assistants, physiotherapists, audiologists, nutritionists, psychologists, occupational therapists and administrative officers), with employment link at the hospital under study who agree to participate by signing an informed consent form are going to be enrolled.

Exclusion Criteria:

The exclusion criteria meet professionals who will be on sick leave, vacation, those who will not to be registered to carry out the intervention and those who will refuse to answer the questionnaire, despite to having shown interest in participating in the lecture and practical class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Mastroianni, PhD, Study Chair — School of Pharmaceutical Sciences of Unesp; Fabiana R Varallo, Master, Principal Investigator — School of Pharmaceutical Sciences of Unesp
Locations (1):
- Hospital Estadual Américo Brasiliense, Américo Brasiliense, São Paulo, Brazil

REFERENCES:
- [Background] Figueiras A, Tato F, Fontainas J, Gestal-Otero JJ. Influence of physicians' attitudes on reporting adverse drug events: a case-control study. Med Care. 1999 Aug;37(8):809-14. doi: 10.1097/00005650-199908000-00010. PMID 10448723
- [Background] Herdeiro MT, Figueiras A, Polonia J, Gestal-Otero JJ. Physicians' attitudes and adverse drug reaction reporting : a case-control study in Portugal. Drug Saf. 2005;28(9):825-33. doi: 10.2165/00002018-200528090-00007. PMID 16119975
- [Background] Herdeiro MT, Figueiras A, Polonia J, Gestal-Otero JJ. Influence of pharmacists' attitudes on adverse drug reaction reporting : a case-control study in Portugal. Drug Saf. 2006;29(4):331-40. doi: 10.2165/00002018-200629040-00004. PMID 16569082
- [Background] Gerritsen R, Faddegon H, Dijkers F, van Grootheest K, van Puijenbroek E. Effectiveness of pharmacovigilance training of general practitioners: a retrospective cohort study in the Netherlands comparing two methods. Drug Saf. 2011 Sep 1;34(9):755-62. doi: 10.2165/11592800-000000000-00000. PMID 21830837
- [Background] Pedros C, Vallano A, Cereza G, Mendoza-Aran G, Agusti A, Aguilera C, Danes I, Vidal X, Arnau JM. An intervention to improve spontaneous adverse drug reaction reporting by hospital physicians: a time series analysis in Spain. Drug Saf. 2009;32(1):77-83. doi: 10.2165/00002018-200932010-00007. PMID 19132807
- [Background] Figueiras A, Herdeiro MT, Polonia J, Gestal-Otero JJ. An educational intervention to improve physician reporting of adverse drug reactions: a cluster-randomized controlled trial. JAMA. 2006 Sep 6;296(9):1086-93. doi: 10.1001/jama.296.9.1086. PMID 16954488
- [Background] Herdeiro MT, Ribeiro-Vaz I, Ferreira M, Polonia J, Falcao A, Figueiras A. Workshop- and telephone-based interventions to improve adverse drug reaction reporting: a cluster-randomized trial in Portugal. Drug Saf. 2012 Aug 1;35(8):655-65. doi: 10.1007/BF03261962. PMID 22788235
- [Background] Herdeiro MT, Polonia J, Gestal-Otero JJ, Figueiras A. Improving the reporting of adverse drug reactions: a cluster-randomized trial among pharmacists in Portugal. Drug Saf. 2008;31(4):335-44. doi: 10.2165/00002018-200831040-00007. PMID 18366244
- [Background] Ribeiro-Vaz I, Herdeiro MT, Polonia J, Figueiras A. Strategies to increase the sensitivity of pharmacovigilance in Portugal. Rev Saude Publica. 2011 Feb;45(1):129-35. doi: 10.1590/s0034-89102010005000050. Epub 2010 Nov 12. English, Portuguese. PMID 21085884
- [Background] Biagi C, Montanaro N, Buccellato E, Roberto G, Vaccheri A, Motola D. Underreporting in pharmacovigilance: an intervention for Italian GPs (Emilia-Romagna region). Eur J Clin Pharmacol. 2013 Feb;69(2):237-44. doi: 10.1007/s00228-012-1321-7. Epub 2012 Jun 17. PMID 22706618

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Post Educational Intervention: Multifaceted educational intervention in pharmacovigilance
  Multifaceted educational intervention: 1- Application of questionnaire of knowledge, attitudes and skills in pharmacovigilance.
  2- Lecture regarding the theoretical framework and importance of pharmacovigilance, and distribution of educational material 3- Distribution of educational material 4- Practical class to explain the correct fill of adverse drug events form 5- Reapplication of questionnaire of knowledge, attitudes and skills in pharmacovigilance.
Period: Overall Study
Arm/Group | Subjects Post Educational Intervention
Started | 203
Completed | 173
Not Completed | 30
Not completed — Did not completed all meetings | 30

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Post Educational Intervention
Number analyzed (Participants) | 173
Age, Continuous [Median (Standard Deviation); unit: years] | 30.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 23
Region of Enrollment [Number; unit: participants]
  Brazil | 173

OUTCOME MEASURES:

1. Primary Outcome: Absolute Number of ADE Reporting (Change Behavior of Health Professionals)
Description: Investigators are going to verify the numbers of adverse drug events reported by health professionals which was made 12 months before educational intervention. A follow up across 12 months post-educational intervention also will be performed, in order to identify the number of adverse drug events reported by health professionals. Prevalence of ADE in both periods will be estimated and compared, in order to asses the impact of the intervention on change behavior of health professionals.
Time Frame: 12 months
Population: Before educational intervention, health professionals reported only three adverse drug events, related to therapeutic failure. However, after the study, the number of reports rise 70-fold, since subjects reported 165 medication errors, 26 adverse drug reactions, 18 quality deviations, 5 therapeutic failure and one off-label use.
Measure: Number; unit: absolute number of adverse drug events
Groups:
- Subjects Prior to Educational Intervention: Number of health professionals who had the potential to report adverse drug reaction, before the educational intervention
Arm/Group | Subjects Post Educational Intervention | Subjects Prior to Educational Intervention
Number analyzed (Participants) | 173 | 173
absolute number of adverse drug events | 215 | 3

2. Secondary Outcome: Knowledge (Awareness) Regarding Pharmacovigilance
Description: Knowledge assessment will be performed by content analysis of answers obtained from questionnaire, being assigned scores from zero to ten. Definitions related to pharmacovigilance of World Health Organization will be considered gold-standard answers. Scores below five will be classified as unsatisfactory, among five and 7.5 were considered regular and above 7.6 satisfactory on the knowledge acquisition.The questionnaire will be applied in the first (prior to educational intervention) and fourth (post-educational intervention period) meetings. Data will be compared, in order to assess the impact of educational intervention on knowledge of health professionals.
Time Frame: Two days
Population: The subjects were assessed regarding pharmacovigilance´s knowledge prior to educational interventions and after as well, in order to evaluate the effectiveness of the study in aware health professionals to report adverse drug events.
Measure: Median (Full Range); unit: percentage of right answers
Groups:
- Subjects Post Educational Intervention: Knowledge of health professionals after multifaceted educational intervention in pharmacovigilance
  Multifaceted educational intervention: 1- Application of questionnaire of knowledge, attitudes and skills in pharmacovigilance.
  2- Lecture regarding the theoretical framework and importance of pharmacovigilance, and distribution of educational material 3- Distribution of educational material 4- Practical class to explain the correct fill of adverse drug events form 5- Reapplication of questionnaire of knowledge, attitudes and skills in pharmacovigilance.
- Subjects Prior to Educational Intervention: Knowledge of health professionals before the educational intervention regarding pharmacovigilance
Arm/Group | Subjects Post Educational Intervention | Subjects Prior to Educational Intervention
Number analyzed (Participants) | 173 | 173
percentage of right answers | 5.2 [0.9 to 9.3] | 2.3 [0.0 to 6.6]
Statistical Analysis 1: Comparison: Subjects Post Educational Intervention; Test type: Superiority or Other; p = 0.00001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Quality of ADE Reports
Description: Skills evaluation will be carried out according to the perception of the voluntary regarding the relevance´s degree of the information to be filled in ADE form. Therefore, in the first (prior to educational intervention) and fourth (post-educational intervention period) meetings, subjects will be asked to highlight the fields of ADE form, according to unnecessary, necessary or essential information to be reported. Minimal and desirable criteria to be filled in ADE form preconized by Pan-American Health Organization will be considered gold-standard answers. Scores from zero to ten will be assigned, according to gold-standard answers. Data will be compared, in order to estimate the impact of educational intervention on skills to fill ADE form.
Time Frame: Two days
Population: The subjects were assessed regarding pharmacovigilance´s skills prior to educational interventions and after as well, in order to evaluate the effectiveness of the study in contribute on the improvement of the quality of information inserted on the form.
Measure: Median (Full Range); unit: percent of correctly filled forms
Groups:
- Subjects Post Educational Intervention: Skills of health professionals in fill correctly the adverse drug events form after multifaceted educational intervention in pharmacovigilance
  Multifaceted educational intervention: 1- Application of questionnaire of knowledge, attitudes and skills in pharmacovigilance.
  2- Lecture regarding the theoretical framework and importance of pharmacovigilance, and distribution of educational material 3- Distribution of educational material 4- Practical class to explain the correct fill of adverse drug events form 5- Reapplication of questionnaire of knowledge, attitudes and skills in pharmacovigilance.
- Subjects Prior to Educational Intervention: Skills of health professionals in fill correctly the adverse drug events form before educational intervention
Arm/Group | Subjects Post Educational Intervention | Subjects Prior to Educational Intervention
Number analyzed (Participants) | 173 | 173
percent of correctly filled forms | 5.2 [0.0 to 9.2] | 3.9 [0.0 to 8.0]
Statistical Analysis 1: Comparison: Subjects Post Educational Intervention; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed.
Description: Adverse Events were not monitored/assessed.
Arm/Group | Subjects Post Educational Intervention
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes